CLINICAL TRIAL: NCT02713425
Title: Pediatric Anxiety Intervention With an Entertaining Video Game: Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Stephen Whiteside, Associate Professor of Psychology, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14-000162
Record Dates: First submitted 2016-03-15; First posted 2016-03-18 (Estimated); Results first posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Anxiety
Keywords: Anxiety; Social Phobia; Separation Anxiety; Generalized Anxiety; GAD; Phobia; video game; teen; youth; child; adolescent
MeSH Terms: conditions — Anxiety Disorders; Phobia, Social; Anxiety, Separation; Generalized Anxiety Disorder; Phobic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm - Entertaining Video Game (Experimental): The children in this study will have a single visit. During this visit they will be introduced to the game. The child will then interact with the game and after they have finished, they will be asked questions about their experience with the game. Parents will observe and provide their own feedback about the game.
  Interventions: Device: Entertaining Video Game

INTERVENTIONS:
Device: Entertaining Video Game — Children between 7 & 17 with a social anxiety disorder will be invited to participate in this study. They will attend a single visit. During the visit they will use the therapeutic game. They will be monitored while using the game. After the completion, they will be asked questions regarding their experience with this therapeutic game.

SUMMARY:
This research study aims to test the feasibility and effectiveness of using an entertaining video game as an addition to traditional therapy for the treatment of anxiety disorders in youth, particularly those youth who may have limited access to mental health treatment in the traditional clinical setting.

DETAILED DESCRIPTION:
The purpose of this research is to learn whether or not youth with social anxiety find a therapeutic video game engaging and useful. Children between the ages of 7 & 17 who have been diagnosed with a social anxiety disorder will be invited to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 7 to 17
2. Primary diagnosis of:

   1. social phobia,
   2. separation anxiety disorder
3. A parent or other primary care giver available to participate with the child in all assessment and treatment activities
4. Estimated average intelligence
5. English speaking
6. Received les than 3 treatment sessions for social anxiety disorder

Exclusion Criteria:

1. History of and/or current diagnosis of:

   1. psychosis,
   2. autism,
   3. bipolar disorder,
   4. mental retardation,
   5. oppositional defiant disorder,
   6. PTSD,
   7. selective mutism, or
   8. major depressive disorder
2. Current suicidality or recent suicidal behavior
3. Parent to be involved in study who is unable to adequately participate due to intellectual or psychiatric difficulties
4. Starting or changing the dosage of a psychiatric medication in the last two months

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Whiteside, Ph.D., L.P., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm - Entertaining Video Game: The children in this study will have a single visit. During this visit they will be introduced to the game. The child will then interact with the game and after they have finished, they will be asked questions about their experience with the game.
  Entertaining Video Game: Children between 7 & 17 with a social anxiety disorder will be invited to participate in this study. They will attend a single visit. During the visit they will use the therapeutic game. They will be monitored while using the game. After the completion, they will be asked questions regarding their experience with this therapeutic game.
Period: Overall Study
Arm/Group | Single Arm - Entertaining Video Game
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: We had a total of 20 children complete the study.
Arm/Group | Single Arm - Entertaining Video Game
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Subjective Units of Distress Scale (SUDS) at End of Session
Description: Subjective Units of Distress Scale (SUDs) - of 0 to 10 ratings, where 0 indicates that they feel no anxiety whatsoever and 10 indicates that they are experiencing maximum distress. The child interacts with the game for up to 30 minutes. The interviewer observes and records the child's interaction with the game. The child then has an opportunity to perform a real life exposure. For the remainder of the time, the interviewer will interview the child about his/her experience with the game. They will also get feedback from the parent.
Time Frame: approximately 10 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm - Entertaining Video Game
Number analyzed (Participants) | 20
score on a scale | 0.74 (2.4)

2. Secondary Outcome: Average Child Rating of Preferring the Game to Not Having the Game
Description: rating of 0(without) to 10 (with) preference to use game
Time Frame: approximately 30 minutes
Population: children with anxiety piloting game
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Arm - Entertaining Video Game
Number analyzed (Participants) | 20
units on a scale | 6.22 (2.6)

ADVERSE EVENTS:
Time Frame: The patients were assessed over an approximately two to three hour period
Description: Participants were monitored during the study for AE/SAE's. None of the patients experienced an AE or SAE. The parent and child has been combined due to the parent having to answer just a couple of questions at the end of the study where as the child participated in the whole study.
Arm/Group | Single Arm - Entertaining Video Game
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-03-14): https://cdn.clinicaltrials.gov/large-docs/25/NCT02713425/SAP_000.pdf
  • Study Protocol (2016-10-04): https://cdn.clinicaltrials.gov/large-docs/25/NCT02713425/Prot_001.pdf